CLINICAL TRIAL: NCT06076980
Title: Haemodynamic Effects of Paracetamol (Acetaminophen) as Extended Intravenous Infusion Versus Intravenous Bolus in Septic Shock Patients
Brief Title: Heamodynamic Effects of Paracetamol in Septic Shock Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ayah Mohammed Khalil (Other)
Responsible Party: Sponsor-Investigator, Ayah Mohammed Khalil, Principal Investigator, Senior clinical pharmacist in Department of Clinical Pharmacy, Cairo University Hospitals (Kasr alainy), Cairo, Egypt., Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: paracetamol in septic shock
Record Dates: First submitted 2023-09-25; First posted 2023-10-11 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Septic Shock; Sepsis
Keywords: acetaminophen; paracetamol; septic shock; hemodynamic effects; blood pressure; icu
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo group (Placebo Comparator): placebo group (100 ml normal saline over 15 minutes)
  Interventions: Drug: Normal saline
- bolus group (Experimental): bolus group (1000mg/100 ml paracetamol over 15 minutes)
  Interventions: Drug: Paracetamol
- Extended infusion group (Experimental): Extended infusion (1000mg/100 ml paracetamol over 3 hours)
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — compare the hemodynamic parameters of paracetamol as bolus versus extended infusion
  Other Names: acetaminophen
  Arms: Extended infusion group; bolus group
Drug: Normal saline — as placebo
  Arms: Placebo group

SUMMARY:
Sepsis is life-threatening organ dysfunction caused by a dysregulated host response to infection. Septic shock is defined as sepsis that has circulatory, cellular, and metabolic abnormalities that are associated with a greater risk of mortality than sepsis alone. Clinically, this includes patients who fulfill the criteria for sepsis who, despite adequate fluid resuscitation, require vasopressors to maintain a mean arterial pressure ≥65 mmHg and have a lactate >2 mmol/L (>18 mg/dL). Feve is a common sign of infection in septic shock critically ill patients. Many critically ill patients experience pain. Paracetamol is considered safe and currently one of the most common antipyretics and used as part of multimodal analgesia for acute pain in the intensive care unit. According to the company's product information leaflet, the rate of hypotension complicating intravenous paracetamol treatment ranges from 0.01 to 0.1%. However, recent studies reported a much higher incidence and may be harmful in critically ill adults. The hemodynamic effects of intravenous (IV) paracetamol are unknown in septic shock patients, that the most vulnerable population and hemodynamically unstable.

The aim of this study is to assess the incidence of hypotension of the extended intravenous paracetamol (acetaminophen) infusion over three hours in comparing with intravenous paracetamol bolus over 15 minutes in hemodynamically unstable patients (septic shock).

DETAILED DESCRIPTION:
Sepsis, inflammatory response to infection, contributes directly or indirectly to mortality in the majority of critically ill patients. An elevated cardiac index and a decreased systemic vascular resistance leading to hypotension and hypoperfusion of vital organs characterize the early stage of septic shock. The hypotensive state is often not amenable to fluid resuscitation alone and requires institution of vasoactive agents to counter the profound fall in systemic vascular resistance, which is an integral feature of septic shock .

Acetaminophen is the antipyretic and analgesic that is most often given to hospitalized patients, including those in critical care units. The mechanism of action of acetaminophen remains incompletely understood, but the antipyretic response appears to be due to blocking cyclooxygenase-II and inhibiting prostaglandin-II synthesis in the central nervous system.

Intravenous (IV) acetaminophen has gained popularity for inpatient management of acute pain for its practical and clinical advantages. IV administration is associated with more predictable pharmacokinetic performance compared with rectal (30%-40% bioavailability) and oral dosage forms of acetaminophen (60%-70% bioavailability).

Predictable kinetics as well as ease of IV administration has made it an especially attractive option in the critically ill patients who have altered gut absorption secondary to numerous pathophysiological and therapeutic influences .

IV acetaminophen has shown promise in improving patient satisfaction, managing fever, and decreasing postoperative opioid requirements. These features have made it one of the most widely ordered medications within critical care and surgical services.

Product information for IV acetaminophen lists mild effects such as nausea or vomiting among the most common adverse events (incidence ≥ 5%), with the estimated incidence of more serious adverse effects such as hypotension being <1%. However, there have been an increasing number of randomized controlled trials which indicated that the incidence of IV acetaminophen-induced hypotension may be higher than previously reported by manufacturers. These publications have prompted investigators to look more closely at the possible untoward effects of IV acetaminophen across a variety of populations. . None of these studies examined whether the extended infusion of IV paracetamol can minimize the degree of hypotension in critically heamodynamic unstable patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age adult ≥ 18 years old.
2. The patient fulfills the criteria of septic shock definition:

   * Sepsis needs vasopressor therapy.
   * Serum lactate level greater than 2 mmol/l (SSC 2016).
3. Patient with contractility greater than 40%

Exclusion Criteria:

1. paracetamol hypersensitivity or allergy.
2. Acute liver injury or failure
3. Childs-Pugh C liver disease
4. Heat stroke.
5. Malignant hyperthermia.
6. Neuroleptic Malignant Syndrome.
7. Continous renal replacement therapy.
8. Ventricular assist device.
9. Around-the-clock scheduled of acetaminophen-containing medications administration or non-steroidal anti-inflammatory drugs.
10. Pregnancy/lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
The incidence of hypotension . | pre intervention and six hours after the intervantion
  defined as a decrease in SBP ≥ 20٪ from baseline, by extended infusion of intravenous paracetamol

SECONDARY OUTCOMES:
The changes in hemodynamic parameters | pre intervention and six hours after the intervantion
  Changes in mean arterial pressure(mmHg), diastolic blood pressure (mmHg)
The changes in hemodynamic parameters | pre intervention and six hours after the intervantion
  Changes in cardiac output ( L/min)
The changes in hemodynamic parameters | pre intervention and six hours after the intervantion
  Changes in heart rate (bpm)
The changes in hemodynamic parameters | pre intervention and six hours after the intervantion
  Changes in central venous pressure (mmHg)
The changes in temperature | pre intervention and six hours after the intervantion
  Changes in temperature (celsius)
The changes in vassopresors and fluid bolus | pre intervention and six hours after the intervantion
  changes in vassopresors infusion rate (mcg/ min) and fluid bolus
The changes in vassopresors and fluid bolus | pre intervention and six hours after the intervantion
  changes in fluid bolus (ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maxwell EN, Johnson B, Cammilleri J, Ferreira JA. Intravenous Acetaminophen-Induced Hypotension: A Review of the Current Literature. Ann Pharmacother. 2019 Oct;53(10):1033-1041. doi: 10.1177/1060028019849716. Epub 2019 May 3. PMID 31046402

DOCUMENTS (1):
  • Study Protocol (2020-08-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT06076980/Prot_000.pdf